CLINICAL TRIAL: NCT01865084
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 3 Trial of Tadalafil for Duchenne Muscular Dystrophy
Brief Title: A Study of Tadalafil for Duchenne Muscular Dystrophy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study is being terminated for lack of efficacy
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15122; H6D-MC-LVJJ (Other: Eli Lilly and Company)
Record Dates: First submitted 2013-05-24; First posted 2013-05-30 (Estimated); Results first posted 2017-03-01 (Actual); Last update posted 2019-10-09 (Actual); Status verified 2019-09

CONDITIONS: Muscular Dystrophy, Duchenne
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — Tadalafil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Experimental): Placebo taken orally once daily.
  Interventions: Drug: Placebo
- 0.3 mg/kg Tadalafil (Experimental): 0.3 milligram per kilogram (mg/kg) tadalafil taken orally once daily.
  Interventions: Drug: Tadalafil
- 0.6 mg/kg Tadalafil (Experimental): 0.6 mg/kg tadalafil taken orally once daily.
  Interventions: Drug: Tadalafil

INTERVENTIONS:
Drug: Tadalafil — Administered orally
  Other Names: LY450190; Cialis
  Arms: 0.3 mg/kg Tadalafil; 0.6 mg/kg Tadalafil
Drug: Placebo
  Other Names: Administered orally
  Arms: Placebo

SUMMARY:
The main purpose of this study is to determine if tadalafil can slow the decline in walking ability of boys who have Duchenne muscular dystrophy (DMD). The study will also assess the safety of tadalafil and any side effects that might be associated with it in boys who have DMD. Participants will receive study treatment (tadalafil or placebo) for the first 48 weeks of the study, and can then continue into an open label extension (OLE) that consists of two periods during which all participants will receive tadalafil. In OLE period 1, all participants will receive tadalafil for 48 weeks. Participants completing OLE period 1 will continue into OLE period 2 and will receive tadalafil for at least another 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Ambulant males with Duchenne muscular dystrophy (DMD) confirmed by typical clinical presentation (onset of clinical signs or symptoms before 6 years of age supported by an elevated serum creatinine kinase level, and ongoing difficulty with walking) together with either a record of a genetic confirmation of the DMD diagnosis, or a record of muscle biopsy showing near-complete dystrophin deficiency (excluding revertant fibers)
* Receiving systemic corticosteroids for a minimum of 6 months immediately prior to screening, with no significant change in total daily dosage or dosing regimen (except those adjusting for weight changes) for a minimum of 3 months immediately prior to screening and a reasonable expectation that total daily dosage and dosing regimen will not change significantly (except for adjustments for weight) for the duration of the study
* Able to complete the six minute walk distance (6MWD) test with results within 20% of each other at a minimum of 2 pre-randomization assessments
* Left ventricular ejection fraction (LVEF) ≥50% as determined by echocardiogram
* Written informed consent from parents/legal guardian will be obtained prior to any study procedure being performed. In addition, the child may be required to give documented assent, if capable.

Exclusion Criteria:

* Symptomatic cardiomyopathy or heart failure
* Change in prophylactic treatment for heart failure within 3 months prior to start of study treatment
* Cardiac rhythm disorder
* History of participation in gene or cell-based therapy , or antisense oligonucleotide or stop codon read-through therapy
* Unable to take orally administered tablets
* Use of any pharmacologic treatment, other than corticosteroids, that might have an effect on muscle strength within 3 months prior to the start of study treatment (for example, growth hormone, anabolic steroids including testosterone)
* New or changed treatment with herbal or dietary supplements being taken with an expectation of an effect on muscle strength or function during 1 month prior to first dose of study drug
* Surgery that might have an effect on muscle strength or function within 3 months before study entry or planned surgery at any time during the study
* Evidence of a lower limb injury that may affect performance on the 6MWD
* Severe behavioral problems, including severe autism or attention deficit disorders, that may interfere with completion of the 6MWD
* Any contraindication to tadalafil (use of any form of organic nitrate, either regularly and/or intermittently, or known serious hypersensitivity to tadalafil)
* History of significant renal insufficiency or clinical evidence of cirrhosis
* Have known allergy to any of the excipients in tadalafil tablets, notably lactose
* Current Phosphodiesterase Type 5 (PDE5) inhibitor therapy or treatment within the past 6 months

Ages: 7 Years to 14 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 331 (Actual)
Dates: Start 2013-09; Primary Completion 2015-12 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (62):
- United States (23):
  - Cedars Sinai Medical Center, Los Angeles, California
  - University of California, Davis - Health Systems, Sacramento, California
  - Children's Hospital, Aurora, Colorado
  - University of Florida Health Science Center, Gainesville, Florida
  - NW Florida Clinical Research Group, Gulf Breeze, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Ann and Robert Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Washington University Medical Center, St Louis, Missouri
  - Carolinas Healthcare System, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Childrens Hospital Medical Center, Cincinnati, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Pennsylvania State University College of Medicine, Hershey, Pennsylvania
  - Childrens Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Childrens Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Children's Medical Center Dallas, Dallas, Texas
  - Univ of Texas Health Science Center at San Antonio, San Antonio, Texas
  - University of Utah School of Medicine, Salt Lake City, Utah
  - Children of the King's Daughters, Norfolk, Virginia
  - Seattle Children's Hospital Research Foundation, Seattle, Washington
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Caba, Argentina
- Belgium (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ghent
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leuven
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Liège
- Canada (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Calgary, Alberta
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vancouver, British Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Winnipeg, Manitoba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Halifax, Nova Scotia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., London, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ottawa, Ontario
- France (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Angers
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nantes
- Germany (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dresden
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Essen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Freiburg im Breisgau
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Göttingen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Munich
- Italy (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Genova
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Milan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Padua
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rome
- Japan (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aichi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nagano
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saitama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo
- Netherlands (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leiden
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nijmegen
- University of Puerto Rico, Medical Sciences Campus, San Juan, Puerto Rico
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Moscow, Russia
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul, South Korea
- Spain (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Donostia / San Sebastian
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Valencia
- Taiwan (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kaohsiung City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taipei
- Turkey (Türkiye) (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Adana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ankara
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Background] McDonald CM, Henricson EK, Han JJ, Abresch RT, Nicorici A, Elfring GL, Atkinson L, Reha A, Hirawat S, Miller LL. The 6-minute walk test as a new outcome measure in Duchenne muscular dystrophy. Muscle Nerve. 2010 Apr;41(4):500-10. doi: 10.1002/mus.21544. PMID 19941337
- [Derived] Cox D, Byrne B, Hammers DW, Landry J, Sweeney HL. Effect of Tadalafil on cardiac function and left ventricular dimensions in Duchenne muscular dystrophy: safety and cardiac MRI substudy results from a randomized, placebo-controlled trial. BMC Cardiovasc Disord. 2025 Apr 11;25(1):276. doi: 10.1186/s12872-025-04727-3. PMID 40217158
- [Derived] Victor RG, Sweeney HL, Finkel R, McDonald CM, Byrne B, Eagle M, Goemans N, Vandenborne K, Dubrovsky AL, Topaloglu H, Miceli MC, Furlong P, Landry J, Elashoff R, Cox D; Tadalafil DMD Study Group. A phase 3 randomized placebo-controlled trial of tadalafil for Duchenne muscular dystrophy. Neurology. 2017 Oct 24;89(17):1811-1820. doi: 10.1212/WNL.0000000000004570. Epub 2017 Sep 29. PMID 28972192

RESULTS

PARTICIPANT FLOW:
Period: Double Blind Period (DB)
Arm/Group | Placebo | 0.3 mg/kg Tadalafil | 0.6 mg/kg Tadalafil
Started | 116 | 102 | 113
Received at Least One Dose of Study Drug | 116 | 102 | 112
Completed | 111 | 98 (One participant stopped therapy during the DB period but remained in the study for follow-up.) | 107
Not Completed | 5 | 4 | 6
Not completed — Adverse Event | 2 | 2 | 1
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Withdrawal by Parent/Guardian | 2 | 2 | 4
Not completed — Withdrawal by Subject | 1 | 0 | 0
Period: Open Label Extension (OLE) Period
Arm/Group | Placebo | 0.3 mg/kg Tadalafil | 0.6 mg/kg Tadalafil
Started | 0 (Participants who were on Placebo during the double blind period were assigned tadalafil during OLE.) | 150 (Participants who were on Placebo during the double blind period were assigned tadalafil during OLE.) | 165 (Participants who were on Placebo during the double blind period were assigned tadalafil during OLE.)
Completed | 0 | 139 | 158
Not Completed | 0 | 11 | 7
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 0 | 2
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Withdrawal by Parent/Guardian | 0 | 8 | 2
Not completed — Withdrawal by Subject | 0 | 2 | 2

BASELINE CHARACTERISTICS:
Population: All participants who were randomized to study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 0.3 mg/kg Tadalafil | 0.6 mg/kg Tadalafil | Total
Number analyzed (Participants) | 116 | 102 | 113 | 331
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.4 (1.76) | 9.9 (2.26) | 9.5 (1.71) | 9.6 (1.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 116 | 102 | 113 | 331
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 2 | 2
  Asian | 15 | 16 | 20 | 51
  Native Hawaiian or Other Pacific Islander | 3 | 1 | 3 | 7
  Black or African American | 0 | 0 | 1 | 1
  White | 96 | 82 | 84 | 262
  More than one race | 2 | 3 | 2 | 7
  Unknown or Not Reported | 0 | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 7 | 4 | 6 | 17
  Russian Federation | 4 | 4 | 4 | 12
  United States | 39 | 34 | 34 | 107
  Japan | 6 | 5 | 6 | 17
  Spain | 9 | 7 | 12 | 28
  Canada | 8 | 7 | 8 | 23
  Netherlands | 2 | 1 | 3 | 6
  Turkey | 5 | 7 | 8 | 20
  Belgium | 8 | 5 | 4 | 17
  Taiwan | 6 | 4 | 8 | 18
  Korea, Republic of | 3 | 4 | 5 | 12
  Italy | 8 | 8 | 8 | 24
  France | 3 | 2 | 2 | 7
  Germany | 8 | 10 | 5 | 23

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Six Minute Walk Distance (6MWD) in Meters
Description: 6MWD measured the distance in meters a participant was able to walk in 6 minutes. The study used 6MWD procedure modified specifically for use in boys with Duchenne muscular dystrophy (DMD), including standardized verbal encouragement at specific intervals to maintain attention to the test, and use of a "safety chaser" to walk behind the participant during testing (McDonald et al., 2010a). The LS mean (LSM) change from baseline, standard error was derived using mixed model repeated measures (MMRM) methodology with factors for pooled country, treatment, visit, treatment-by-visit interaction and baseline 6MWD as a covariate.
Time Frame: Baseline, Week 48
Population: All randomized participants who received at least one dose of study drug who had a baseline and at least one post-baseline measurement.
Measure: Least Squares Mean (Standard Error); unit: Meters
Groups:
- 0.3 mg/kg Tadalafil: 0.3 mg/kg tadalafil taken orally once daily.
- 0.6 mg/kg Tadalafil: 0.6 mg/kg taken tadalafil orally once daily.
Arm/Group | Placebo | 0.3 mg/kg Tadalafil | 0.6 mg/kg Tadalafil
Number analyzed (Participants) | 113 | 101 | 111
Meters | -50.99 (9.316) | -64.71 (9.809) | -59.08 (9.397)
Statistical Analysis 1: Comparison: Placebo vs 0.3 mg/kg Tadalafil; Test type: Superiority or Other; p = 0.307, Mixed Models Analysis — The p-value is based on the treatment difference LS Mean changes from baseline between tadalafil and placebo
Statistical Analysis 2: Comparison: Placebo vs 0.6 mg/kg Tadalafil; Test type: Superiority or Other; p = 0.538, Mixed Models Analysis — The p-value is based on the treatment difference LS Mean changes from baseline between tadalafil and placebo

2. Secondary Outcome: Change From Baseline in the North Star Ambulatory Assessment (NSAA) Global Score
Description: The NSAA is a functional scale specifically designed for ambulant boys with DMD that can provide additional information on motor functions important in maintaining normal ambulation and other activities important to everyday life. The NSAA is a 17-item evaluation of standing, ability to transition from lying to sitting, sitting to standing, and other mobility assessments. Each of the 17 items is evaluated on an ordinal scale of 0, 1, or 2, with higher scores reflecting better performance on the assessment, for a total maximum score of 34. This score was transformed to a 0 to 100 scale for the key analysis (referred to as linearized), with higher transformed scores reflecting better performance.The LS mean (LSM) change from baseline standard error was derived using mixed model repeated measures methodology (MMRM) with factors for pooled country, treatment, visit, treatment-by-visit interaction and Day 1 value as baseline covariate.
Time Frame: Baseline, Week 48
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | 0.3 mg/kg Tadalafil | 0.6 mg/kg Tadalafil
Number analyzed (Participants) | 116 | 102 | 112
Units on a scale | -8.80 (1.104) | -9.31 (1.181) | -8.96 (1.115)

3. Secondary Outcome: Change From Baseline in Timed Function Tests in Seconds
Description: Timed function tests included time it took to rise from floor, walk 10 meters, ascend 4 stairs, and descend 4 stairs.The lower the time in seconds taken, the better the performance. The LS mean change from baseline, standard error, was derived using mixed model repeated measures methodology (MMRM) with factors for pooled country, treatment, visit, treatment-by-visit interaction and Day 1 value as baseline covariate.
Time Frame: Baseline, Week 48
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Seconds
Arm/Group | Placebo | 0.3 mg/kg Tadalafil | 0.6 mg/kg Tadalafil
Number analyzed (Participants) | 116 | 96 | 110
Seconds
  Rise from the Floor(n=92,75,89) | 4.16 (1.120) | 3.60 (1.223) | 4.81 (1.156)
  10 Meter Walk/Run(n=105,90,100) | 1.11 (0.204) | 0.95 (0.226) | 1.12 (0.217)
  Stair Climb (n=116,96,110) | 3.96 (1.041) | 4.10 (1.154) | 5.82 (1.072)
  Stair Descend(n=115,95,110) | 3.19 (0.827) | 2.07 (0.915) | 3.27 (0.853)

4. Secondary Outcome: Time to Persistent 10% Worsening in 6MWD
Description: Time on study until the 6MWD becomes 10% less than the baseline 6MWD and continues at that level or lower until the end of study.
Time Frame: Baseline through Week 48
Population: All randomized participants who received at least one dose of study drug who had complete evaluable data. Complete evaluable data was defined as having baseline measurement, complete dates at evaluable visits and a post-baseline measurement at each evaluable visit. Censored participants: placebo=71, 0.3 mg/kg=63, 0.6 mg/kg=61.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Placebo | 0.3 mg/kg Tadalafil | 0.6 mg/kg Tadalafil
Number analyzed (Participants) | 115 | 101 | 111
Days | NA [NA to NA] — These statistics were not estimable due to large number of participants who were censored. | NA [NA to NA] — These statistics were not estimable due to large number of participants who were censored. | NA [NA to NA] — These statistics were not estimable due to large number of participants who were censored.

5. Secondary Outcome: Time to Persistent 10% Worsening in Timed Function Tests (TFT)
Description: Time on study until the TFT becomes 10% worse than the baseline TFT and continues at that level or lower until the end of study. The time to persistent 10% worsening is the observed time after baseline until the first observed timepoint where their time used for the TFTs is >110% of the baseline time and all the time values observed afterward are also >110% of baseline. If the participant discontinues prior to experiencing persistent worsening, this outcome for the participant is censored at the date of discontinuation of the double-blind period.
  Only participants with complete evaluable data were analyzed. Complete evaluable data was defined as having baseline measurement, complete dates at evaluable visits and a post-baseline measurement at each evaluable visit.
Time Frame: Baseline through Week 48
Population: All randomized participants who received at least 1 dose of study drug who had complete evaluable data.Censored participants:Rise from Floor;placebo(pl)=40,0.3 mg/kg=39,0.6 mg/kg=43;Stair Climb;pl=55,0.3 mg/kg=45,0.6 mg/kg=52;10 Meter Walk/Run pl=61,0.3 mg/kg=65,0.6 mg/kg=58,Stair Descend;pl=63,0.3 mg/kg=60,0.6 mg/kg=59.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Placebo | 0.3 mg/kg Tadalafil | 0.6 mg/kg Tadalafil
Number analyzed (Participants) | 116 | 102 | 113
Days
  Rise from the Floor (n=81,67,77) | 253.0 [170.0 to NA] — These statistics were not estimable due to large number of participants who were censored. | NA [NA to NA] — These statistics were not estimable due to large number of participants who were censored. | NA [NA to NA] — These statistics were not estimable due to large number of participants who were censored.
  Stair Climb (n=112,91,107) | 255.0 [252.0 to NA] — These statistics were not estimable due to large number of participants who were censored. | 259.0 [176.0 to NA] — These statistics were not estimable due to large number of participants who were censored. | 253.0 [185.0 to NA] — These statistics were not estimable due to large number of participants who were censored.
  10 Meter Walk/Run (n=98,83,91) | NA [NA to NA] — These statistics were not estimable due to large number of participants who were censored. | NA [NA to NA] — These statistics were not estimable due to large number of participants who were censored. | NA [NA to NA] — These statistics were not estimable due to large number of participants who were censored.
  Stair Descend (n=110,91,108) | NA [NA to NA] — These statistics were not estimable due to large number of participants who were censored. | NA [NA to NA] — These statistics were not estimable due to large number of participants who were censored. | NA [NA to NA] — These statistics were not estimable due to large number of participants who were censored.

6. Secondary Outcome: Change From Baseline in Pediatric Outcomes Data Collection Instrument (PODCI) Scores
Description: PODCI includes a Global Functioning Scale and 5 core scales:Upper Extremity and Physical Function,Transfer/Basic Mobility, Sports/Physical Functioning, Pain/Comfort,and Happiness.The Global Functioning Scale is the mean of the mean scores from 4 of the 5 core scales (all except the happiness core scale).The following PODCI scores were prespecified in the protocol for analysis: Global Functioning, Upper Extremity and Physical Function,Transfer/Basic Mobility, and Sports/Physical Functioning. The Global Functioning Scale and each of the core scales were standardized so that a score of "0" represents a poor outcome/worse health, while "100" is the best possible outcome/best health (i.e., complete range of each score is 0 to 100, with higher scores representing better functioning). The LS mean (LSM) change from baseline,standard error was derived using MMRM with factors for pooled country, treatment, visit, treatment-by-visit interaction and baseline PODC scale as covariate.
Time Frame: Baseline, Week 48
Population: All randomized participants who received at least one dose of study drug who had a baseline and at least one post-baseline measurement. The reason the number of participants analyzed is significantly less than the total number of randomized participants is because PODCI was administered only in English.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | 0.3 mg/kg Tadalafil | 0.6 mg/kg Tadalafil
Number analyzed (Participants) | 41 | 35 | 34
Units on a scale
  Global Functioning Scale (n=41,34,34) | -8.81 (1.770) | -7.36 (1.929) | -7.34 (1.888)
  Upper Extremity & Physical Function | -5.47 (1.901) | -3.73 (2.060) | -2.47 (2.042)
  Transfer/Basic Mobility Core Scale | -14.26 (3.037) | -12.50 (3.260) | -12.78 (3.279)
  Sports/Physical Functioning Core Scale | -12.47 (2.362) | -11.98 (2.552) | -7.88 (2.537)

7. Secondary Outcome: Pharmacokinetics (PK): Apparent Clearance (CL/F) of Tadalafil
Description: The data reported are population estimate and inter-patient variability.
Time Frame: Weeks 4, 12, 24 and 36: -1 Hour up to 24 Hours Postdose
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour (L/hr)
Groups:
- 0.3 mg/kg Tadalafil and 0.6 mg/kg Tadalafil: 0.3 mg/kg tadalafil taken orally once daily.
  0.6 mg/kg tadalafil taken orally once daily.
Arm/Group | 0.3 mg/kg Tadalafil and 0.6 mg/kg Tadalafil
Number analyzed (Participants) | 210
Liter per hour (L/hr) | 1.79 (29.6)

ADVERSE EVENTS:
Description: All randomized participants who received at least one dose of study drug for Placebo - DB, 0.3 mg/kg Tadalafil -DB and 0.6 mg/kg Tadalafil - DB arms during the DB period.
  All randomized participants who received at least one dose of study drug for 0.3 mg/kg Tadalafil - OLE and 0.6 mg/kg Tadalafil - OLE arms during the OLE period.
Groups:
- Placebo - DB: Placebo taken orally once daily.
- 0.3 mg/kg Tadalafil -DB: 0.3 milligram per kilogram (mg/kg) tadalafil taken orally once daily.
- 0.6 mg/kg Tadalafil - DB; 0.6 mg/kg Tadalafil - OLE: 0.6 mg/kg tadalafil taken orally once daily.
- 0.3 mg/kg Tadalafil - OLE: 0.3 mg/kg tadalafil taken orally once daily.
Arm/Group | Placebo - DB | 0.3 mg/kg Tadalafil -DB | 0.6 mg/kg Tadalafil - DB | 0.3 mg/kg Tadalafil - OLE | 0.6 mg/kg Tadalafil - OLE
Serious Adverse Events (participants affected / at risk) | 5/116 | 4/102 | 6/112 | 6/150 | 9/165
Other Adverse Events (participants affected / at risk) | 83/116 | 82/102 | 92/112 | 68/150 | 84/165
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo - DB (N=116) | 0.3 mg/kg Tadalafil -DB (N=102) | 0.6 mg/kg Tadalafil - DB (N=112) | 0.3 mg/kg Tadalafil - OLE (N=150) | 0.6 mg/kg Tadalafil - OLE (N=165)
Myocarditis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abasia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngotonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pneumonia adenoviral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Varicella (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tendinous contracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Extrapyramidal disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Self injurious behaviour (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo - DB (N=116) | 0.3 mg/kg Tadalafil -DB (N=102) | 0.6 mg/kg Tadalafil - DB (N=112) | 0.3 mg/kg Tadalafil - OLE (N=150) | 0.6 mg/kg Tadalafil - OLE (N=165)
Abdominal pain (Gastrointestinal disorders) | 6 (7) | 4 (4) | 9 (9) | 2 (2) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 7 (7) | 5 (6) | 8 (8) | 4 (5) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 10 (10) | 6 (9) | 10 (19) | 9 (13) | 7 (7)
Nausea (Gastrointestinal disorders) | 2 (2) | 7 (8) | 3 (3) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 14 (20) | 6 (6) | 17 (25) | 9 (12) | 10 (11)
Abasia (General disorders) | 6 (6) | 14 (14) | 9 (9) | 12 (12) | 16 (16)
Pyrexia (General disorders) | 4 (4) | 11 (11) | 9 (10) | 7 (8) | 6 (6)
Gastroenteritis (Infections and infestations) | 6 (6) | 4 (4) | 3 (3) | 3 (3) | 2 (2)
Influenza (Infections and infestations) | 9 (9) | 8 (9) | 5 (5) | 3 (3) | 2 (2)
Nasopharyngitis (Infections and infestations) | 16 (26) | 8 (10) | 18 (24) | 8 (10) | 12 (12)
Sinusitis (Infections and infestations) | 6 (11) | 4 (5) | 3 (3) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 10 (18) | 10 (21) | 12 (16) | 6 (15) | 8 (10)
Fall (Injury, poisoning and procedural complications) | 24 (41) | 18 (30) | 22 (41) | 16 (22) | 15 (18)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (15) | 11 (12) | 7 (7) | 7 (7) | 9 (9)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7 (9) | 3 (3) | 3 (4) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 (14) | 6 (6) | 10 (11) | 2 (2) | 4 (4)
Headache (Nervous system disorders) | 36 (92) | 40 (57) | 43 (68) | 8 (12) | 14 (19)
Erection increased (Reproductive system and breast disorders) | 3 (3) | 10 (11) | 17 (18) | 2 (2) | 4 (4)
Spontaneous penile erection (Reproductive system and breast disorders) | 4 (6) | 13 (13) | 13 (14) | 3 (3) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (11) | 4 (4) | 5 (5) | 4 (5) | 5 (5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 (11) | 10 (15) | 6 (8) | 4 (6) | 3 (5)
Rash (Skin and subcutaneous tissue disorders) | 7 (7) | 3 (3) | 5 (5) | 3 (3) | 1 (1)
Flushing (Vascular disorders) | 3 (3) | 8 (8) | 8 (9) | 2 (2) | 2 (2)

LIMITATIONS AND CAVEATS:
The Sponsor concluded that the efficacy results do not provide sufficient justification for continuance of the open-label extension (OLE) period of the study, where all participants were receiving daily treatment with tadalafil.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days